CLINICAL TRIAL: NCT04547582
Title: Spinal Cord Stimulation for Restoration of Function in Lower-Limb Amputees, 90-Day
Acronym: SCS-90
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Additional participants were not enrolled after multiple years of recruitment efforts. Funding expired.
Sponsor: Lee Fisher, PhD (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Lee Fisher, PhD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19010019; 1UH3NS100541-01A1 (NIH)
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Amputation of Lower Extremity; Phantom Limb Pain
Keywords: Phantom Limb Pain; Lower-Limb Amputation; electrodes; stimulation; BKA; pain; sensation
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Spinal cord stimulation (Experimental): Spinal cord stimulator leads (2-3 leads) will be placed in the lumbar epidural space of lower limb amputees to determine if the patient experiences any pain reduction from spinal cord stimulation.
  Participants in this study receive spinal cord stimulation will be trans-tibial amputees that are at least six month post--amputation. Subjects will have varying levels of phantom limb sensation and pain, but should have no other significant neurological disorders.
  Interventions: Device: Spinal cord stimulator

INTERVENTIONS:
Device: Spinal cord stimulator — Spinal cord stimulator leads (2-3 leads) will be placed in the lumbar epidural space of lower limb amputees to determine if the patient experiences any pain reduction from spinal cord stimulation.

SUMMARY:
The goals of this study are to provide sensory information to amputees and reduce phantom limb pain via electrical stimulation of the lumbar spinal cord and spinal nerves. The spinal nerves convey sensory information from peripheral nerves to higher order centers in the brain. These structures still remain intact after amputation and electrical stimulation of the dorsal spinal nerves in individuals with intact limbs and amputees has been demonstrated to generate paresthetic sensory percepts referred to portions of the distal limb. Further, there is recent evidence that careful modulation of stimulation parameters can convert paresthetic sensations to more naturalistic ones when stimulating peripheral nerves in amputees. However, it is currently unclear whether it is possible to achieve this same conversion when stimulating the spinal nerves, and if those naturalistic sensations can have positive effects on phantom limb pain. As a first step towards those goals, in this study, the investigators will quantify the sensations generated by electrical stimulation of the spinal nerves, study the relationship between stimulation parameters and the quality of those sensations, measure changes in control of a prosthesis with sensory stimulation, and quantify the effects of that stimulation on the perception of the phantom limb and any associated pain.

DETAILED DESCRIPTION:
During the study, FDA-cleared spinal cord stimulator leads will be placed in the lumbar epidural space of lower limb amputees and steered laterally towards the dorsal spinal roots under fluoroscopic guidance. This approach is essentially identical to the FDA-cleared procedure in which these devices are placed in the lumbar epidural space for treatment of intractable low back and leg pain. In that procedure, it is common clinical practice to place 2-3 leads temporarily in the epidural space through a percutaneous approach and perform a multiday trial to determine if the patient experiences any pain reduction from spinal cord stimulation. Following the trial, the percutaneous leads are surgically removed, and the patient is referred to a neurosurgeon for permanent surgical implantation.

Similarly, in this study, the device will be tunneled percutaneously through the skin and anchored in place. Using the stylet included with the spinal cord stimulator leads, the devices will be steered laterally under fluoroscopic guidance to target the dorsal spinal nerves. During lab experiments, the leads will be connected to an external stimulator. In this study, the devices will remain in the epidural space for up to 90 days and will be surgically removed. Throughout the study, the investigators will perform a series of psychophysical evaluations to characterize the sensory percepts evoked by epidural stimulation, along with functional evaluations of the effects of stimulation on the ability to control a prosthetic limb. In addition, the investigators will perform surveys to characterize changes in phantom limb sensation and pain that occur during stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have an amputation of one lower limb, at a level between the ankle and knee joints. Minor amputation of the contralateral limb (i.e. toes or partial foot) is not exclusionary.
2. Subjects must be over 6 months post-amputation at the time of lead placement.
3. Subjects must be between the ages of 22 and 70 years old. Participants outside this age range may be at an increased medical risk and have an increased risk of fatigue during testing.
4. Subjects must have used their current prosthesis for at least 6 months and achieved at least K-1 ambulator status at the time of lead placement, as determined by the Amputee Mobility Predictor.

Exclusion Criteria:

1. Subjects must not have any serious disease or disorder that could affect their ability to participate in this study.
2. Female subjects of childbearing age must not be pregnant or breast-feeding.
3. Subjects must not be receiving medications that affect blood coagulation.
4. Subjects must not have an allergy to contrast medium or renal failure that could be exacerbated by the contrast agent used in MRIs. For this study, renal insufficiency will be determined through blood work and defined as BUN of 30 or less and Creatinine of 1.5 or less.
5. Subjects may not have a hemoglobin A1c level above 8.0 mg/dl at time of implant.
6. Subjects may not have any implanted medical devices that are not cleared for MRI.
7. Subjects with a T-Score higher than 63 on the 18-question Brief Symptoms Inventory (BSI-18) who have undergone discussions with and been deemed unsuitable by the Principal Investigator, a study physician, and a psychologist
8. Subjects may not have a cardiac pacemaker.
9. Subjects may not have a cardioverter defibrillator.
10. Subjects may not be currently receiving diathermy therapy.
11. Subjects may not have an implanted infusion pump.
12. Subjects may not be immunosuppressed or currently receiving immunosuppressive medications.
13. Subjects may not have a profession (e.g. radiology technologist) or medical condition (e.g. remissory cancer involved regular follow-up x-rays) that would increase radiation exposure in the 12 months prior to starting or after ending participation in the study.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee E Fisher, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share data with researchers at other centers for the purpose of data analysis and collaboration.
Supporting Information: SAP, ICF
Time Frame: Data will be shared according to guidelines in data sharing agreements.
Access Criteria: We will share with our sponsor and collaborators.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 2021 to 2023 from affiliated amputee clinics. Recruitment continued through 2025, but no additional subjects were enrolled.
Pre-assignment Details: Enrollment is defined as completing informed consent.
Groups:
- Spinal Cord Stimulation: Spinal cord stimulator leads (2-3 leads) will be placed in the lumbar epidural space of lower limb amputees to determine if the patient experiences any pain reduction from spinal cord stimulation.
  Participants in this study receive spinal cord stimulation will be trans-tibial amputees that are at least six month post--amputation. Subjects will have varying levels of phantom limb sensation and pain, but should have no other significant neurological disorders.
  Spinal cord stimulator: Spinal cord stimulator leads (2-3 leads) will be placed in the lumbar epidural space of lower limb amputees to determine if the patient experiences any pain reduction from spinal cord stimulation.
Period: Overall Study
Arm/Group | Spinal Cord Stimulation
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Serious Device-related Adverse Events up to 90 Days Following Implantation
Description: Investigators will track the number of participants experiencing serious device-related adverse events, such as unresolved superficial infection resulting in lead removal, deep infection, inpatient hospitalization, withdrawal from the study due to worsening pain or intolerable dysesthesia, or fracture due to falls related to the study interventions, that occur during the course of and up to 90 days following implantation.
Time Frame: 90 days
Population: One participant was implanted with spinal cord stimulation leads.
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal cord stimulation
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Minimum Amplitude of Pulse Required to Evoke Sensory Percepts
Description: Quantify the threshold stimulus required to evoke sensory percepts during epidural spinal nerve stimulation.
Time Frame: 90 days
Measure: Number; unit: milliamps
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 1
milliamps | 2

3. Primary Outcome: Minimum Charge Required to Evoke a Neurophysiological Response
Description: Quantify the threshold (minimum charge) stimulus required to evoke neurophysiological responses during epidural spinal nerve stimulation
Time Frame: 90 days
Measure: Number; unit: uC (microcoulombs)
Arm/Group | Spinal cord stimulation
Number analyzed (Participants) | 1
uC (microcoulombs) | 1.23

4. Primary Outcome: Location of Evoked Sensation - Missing Toes
Description: Participants reporting sensation on missing toes from spinal cord stimulation.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 1
Participants | 1

5. Primary Outcome: Location of Evoked Sensation - Plantar Surface of Missing Foot
Description: Participants perceiving sensation on the plantar surface of missing foot
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 1
Participants | 1

6. Secondary Outcome: Change in Phantom Limb Pain Using the McGill Pain Questionnaire
Description: The McGill Pain Questionnaire is a questionnaire used to evaluate the severity of pain experienced by the participant. The questionnaire is scaled, with a minimum and maximum pain score of 0 and 78, respectively. The higher the score on the questionnaire, the more intense the pain felt by the participant. A lower score than previously reported represents a decrease in experienced phantom limb pain.
  Before placement of the spinal cord stimulator leads, investigators will document the subject's description of their history of perceived phantom limb. Investigators will ask them to periodically update their perception of the limb throughout experimental sessions, as well as within a month after the device has been removed.
Time Frame: Pre-implant (baseline), Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and post-explant (90 days)
Measure: Number; unit: score on a scale
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 1
score on a scale
  Pre-implant (baseline) | 48
  Week 1 (after implant) | 32
  Week 2 | 45
  Week 3 | 45
  Week 4 | 23
  Week 5 | 38
  Week 6 | 32
  Week 7 | 34
  Week 8 | 17
  Week 9 | 46
  Week 10 | 41
  Week 11 | 65
  Post-explant (90 days) | 47

7. Secondary Outcome: Qualitative Self-report of Evoked Sensations
Description: Document the subjective perception of lumbosacral epidural spinal nerve stimulation for restoration of sensation. The investigators will ask each subject to provide subjective feedback on their perceived utility of the sensory feedback provided by the device. A total of 13 natural descriptors and 5 paresthetic descriptors were presented to participants weekly to describe the sensation provided via spinal cord stimulation. The goal of the study is to elicit more natural than paresthetic descriptors from participants.
  Natural: pressure, tickle, flutter, warm, sharp, prick, cool, pulsing, vibration, itch, urge to move, touch, tap Parethetic: buzz, tingle, shock, electric current, numb
Time Frame: 90 days
Population: For all reported sensations, each electrode was stimulated with a 1-second long pulse train.
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 1
Participants
  More natural than paresthetic descriptors. | 1
  More paresthetic than natural descriptors. | 0

8. Secondary Outcome: Able to Use a Prosthetic Limb With Neural Signals
Description: Investigators will test the subject's success rate during control of prosthetic limb with and without sensory feedback provided by electrical stimulation of the spinal roots. Using either a virtual prosthetic limb or an instrumented prosthesis, stimulation of the spinal roots will be modulated based on signals recorded from the limb.
Time Frame: 90 days
Population: Individuals implanted with spinal cord stimulator leads in lumbar spine
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Cord Stimulation
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 90 days
Description: Self-report by participant
Arm/Group | Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Cord Stimulation (N=1)
Incision pain (Surgical and medical procedures) | 1 (1) — Incision pain following implant
Chest pain after surgery (Surgical and medical procedures) | 1 (1) — Left-sided chest pain after explant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04547582/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04547582/ICF_001.pdf